CLINICAL TRIAL: NCT00775567
Title: Colonic Microbial and Clinical Adaptation to Large Doses of Fructose
Brief Title: Effect of Fructose on Colonic Microflora
Acronym: MEF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Andrew Szilagyi, SMBD Jewish General Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 07111
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2009-02

CONDITIONS: Healthy
Keywords: Fructose; Intolerance; Adaptation; Prebiotic; Healthy men or women 18-40

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): 30g fructose dissolved in water twice a day
  Interventions: Dietary Supplement: Fructose powder
- No Intervention (No Intervention)

INTERVENTIONS:
Dietary Supplement: Fructose powder — 30g in 250ml water twice a day
  Arms: 1

SUMMARY:
Fructose is the principal carbohydrate in fruits and is added to many food products. This 6 carbon sugar is associated with a number of ill effects, like promotion of high triglycerides,precipitation of gout in men,possible depression in women and symptoms of intolerance in a non ethnic dose dependent fashion.However, high fruit and vegetable intake is associated with some epidemiologic evidence in prevention of some cancers like stomach and colorectum.The principal protectors in these products are thought to be antioxidants and other protective chemicals like polyphenols.In addition long chain polymers of fructose:inulin are thought to help protect against cancer through prebiotic effects. In fact poly-fructose molecules are used as prebiotic food supplements and are promoted as aids for a healthy intestine with "balanced microflora".

Polyfructose prebiotics induce some gastrointestinal symptoms of cramps gas bloating and sometimes diarrhea.To date repeated consumption of these polyfructose molecules have not been shown to induce colonic adaptation. Nor is there evidence that fructose intolerant people "adapt " to prolonged ingestion.

These findings are in contrast to findings with lactose intolerance where prolonged ingestion leads to both symptomatic and physiological adaptation.In this interventional study we evaluate whether fructose intolerant people can adapt to moderate dose daily fructose ingestion.The desired outcome is symptomatic, physiological and colonic microfloral adaptation. A failure to detect an increase in bifidobacteria on retesting may suggest that in humans like in some other mammals GLUT5 fructose transport could be induced.

DETAILED DESCRIPTION:
The concept of Colonic Adaptation(CA) to regular carbohydrates has been linked mainly to lactose disaccharide(galactose,glucose) and lactulose(galactose, fructose), a manufactured derivative of lactose. CA is achieved in both cases by short term regular consumption of the targeted sugar which is not digested by the host. The clinical definition of CA includes a measured change in breath hydrogen, reduction of clinical symptoms (Bloat, gas, cramps and at times diarrhea) and an associated increase of bacterial lactase(β-galactosidase. The putative mechanism is through bacterial action which results in enhanced metabolism or expanded bacterial population of specific genus and species of bacteria. The act of CA may incur health benefits through physicochemical changes and especially promotion of health promoting bacteria.

Maldigestion of fructose occurs in the population probably in a dose dependent fashion. The sugar content overwhelms the principal GLUT5 intestinal carrier. In the presence of glucose this non energy dependent system works better(11). In a previous publication we found that the pre test graded ingestion of fructose had no impact on test results. These results were dramatically different from that found for pretest lactose ingestion. The investigators interpreted the results from the fructose study as being consistent with a failure to show CA to regular fructose consumption.

More recently Rao et al however, showed that there may be a threshold level of intake beyond which fructose maldigestion may rapidly increase. This value was thought to be 15-20g. In the case of lactose this was 10g(15). Since in both our studies we used the same dose response analysis(<10,11-19, and >20g/d), it is possible that fructose consuming individuals might not have spilt adequate quantities of fructose into the colon to properly induce and maintain CA. Moreover, there is to our knowledge no information on a possible prebiotic effect of the monosaccharide fructose. Since polymers of fructose are very good prebiotics it may be of interest to determine whether this sugar is capable of prebiotic function in its own right.

The investigators propose to carry out a short term study on 20-30 healthy participants to determine whether a 2 week period of fructose consumption alters clinical CA and intestinal microflora.

Study Outline After an overnight fast, except for water(ad libitum), participants present themselves to the GI lab around 9 am. A 50 gm fructose solution (this dose is associated with a 65% chance of maldigestion(14))will be administered. Breath hydrogen and symptoms will be recorded for 4.5 Hrs at ½ hr intervals. Participants will be asked to fill out a short 3 day diet recall questionnaire targeting fructose ingestion.

Participants will be asked to consume 30g fructose in 150ml of water (lemon juice may be added) twice a day for 14 days.They will then return for a repeat50 g fructose challenge. A small stool sample will be asked from participants at each test period.Another similar group will undergo the same tests but without taking intervening fructose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants

Exclusion Criteria:

* Antibiotics 90 days pre entry
* Use of gastrointestinal motility drugs eg loperamide, metoclopramide significant fiber supplements
* Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Statistically significant reduction in total sum breath hydrogen upon a 50g fructose challenge test. | intervention for 2 weeks per participant

SECONDARY OUTCOMES:
A log 1 change in fecal bifidobacteria or lactobacilli species. | stools retested 2 weeks apart

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Szilagyi, MD, Principal Investigator — SMBD Jewish General Hospital, McGill university School of Medicine
Locations (1):
- SMBD Jewish General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] Szilagyi A, Malolepszy P, Yesovitch S, Vinokuroff C, Nathwani U, Cohen A, Xue X. Fructose malabsorption may be gender dependent and fails to show compensation by colonic adaptation. Dig Dis Sci. 2007 Nov;52(11):2999-3004. doi: 10.1007/s10620-006-9652-9. Epub 2007 Mar 15. PMID 17357833
- [Background] Rao SS, Attaluri A, Anderson L, Stumbo P. Ability of the normal human small intestine to absorb fructose: evaluation by breath testing. Clin Gastroenterol Hepatol. 2007 Aug;5(8):959-63. doi: 10.1016/j.cgh.2007.04.008. Epub 2007 Jul 10. PMID 17625977
- [Background] Szilagyi A, Malolepszy P, Yesovitch S, Nathwani U, Vinokuroff C, Cohen A, Xue X. Inverse dose effect of pretest dietary lactose intake on breath hydrogen results and symptoms in lactase nonpersistent subjects. Dig Dis Sci. 2005 Nov;50(11):2178-82. doi: 10.1007/s10620-005-3028-4. PMID 16240236
- [Background] Briet F, Achour L, Flourie B, Beaugerie L, Pellier P, Franchisseur C, Bornet F, Rambaud JC. Symptomatic response to varying levels of fructo-oligosaccharides consumed occasionally or regularly. Eur J Clin Nutr. 1995 Jul;49(7):501-7. PMID 7588500
- See also: Full article on line — http://www.pagepress.org/gi